CLINICAL TRIAL: NCT07403149
Title: Evaluating the Improvement of Stepping Quality by Using Adapted Shoes
Brief Title: Improving STEP in Stroke Patients
Acronym: I-STEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Maison LLAFIA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP250627; 2025-A01226-43 (Other: ANSM)
Record Dates: First submitted 2025-09-23; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Hemiplegia Following Ischemic Stroke; Disability Physical; Spasticity as Sequela of Stroke; Gluteus Maximus Muscle Atrophy; Equinovarus Foot
Keywords: Stroke; Hemiplegia; equinovarus; orthopedic shoes; REMARCHE® shoes; Walking performance
MeSH Terms: conditions — Stroke; Hemiplegia; Clubfoot

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMARCHE® shoes (Experimental): REMARCHE™ shoes are custom-hand-made, with soles adapted to posture, integrated elevator splint, and raise of the tip of the shoes, and contra-lateral leg elevation to avoid friction of the tip of the ipsilateral foot
  Interventions: Device: REMARCHE® shoes
- Sham REMARCHE® shoes (Sham Comparator): Sham REMARCHE® shoes, custom-hand-made conventional shoes, with same appearance.
  Interventions: Device: Sham REMARCHE® shoes

INTERVENTIONS:
Device: REMARCHE® shoes — REMARCHE® shoes custom-hand-made, with soles adapted to posture, integrated elevator splint, and raise of the tip of the shoes, and contra-lateral leg elevation to avoid friction of the tip of the ipsilateral foot
  Arms: REMARCHE® shoes
Device: Sham REMARCHE® shoes — Sham REMARCHE® shoes, custom-hand-made conventional shoes, with same appearance
  Arms: Sham REMARCHE® shoes

SUMMARY:
Stroke is the leading cause of acquired disability in adults. Stroke causes death in 10% of patients, disability and functional handicap in 60% of cases. Sequelea of hemiplegia include spasticity resulting in great difficulty and slowness in walking, gait instability, increasing the risk of falls.

Deambulation may need help (cane, crutch, tripod cane, walker). Lower limb spasticity includes hypertonia of extensors (gluteus maximus, quadriceps, posterior gastrocnemius) resulting in equinovarus. A neurology deficit may be present on ipsilateral lower limb flexors. Hence the patient walks with rubbing of the tip of the foot (tip-toeing gait), resulting in a "mowing wheatslike" movement of the leg as described in the French literature. Walking is then slowed down, unstable, with increased risk of falls.

In post stroke, during the period of rehabilitation and beyond, it is advisable to wear sports shoes although custom-made shoes improve walking and are reimbursed by the French social security system after prior agreement. Most of patients only wear conventional shoes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18 years
2. With health insurance card " carte vitale " (being affiliated to the French security system) on "ALD" (Affection de longue durée) meaning reimbursement at a 100% rate
3. With a past history of stroke (ischemic or hemorrhagic) with a Rankin score 2 to 4, once stabilized (no more improvement), at least 6 months after stroke onset
4. Spasticity on one side of the body, with spastic walking, with tip-toeing gait, resulting in a "mowing wheats-like" movement of the leg as described in the French literature
5. Patient had full medical examination prior to this research
6. Informed and written consent of the participant.

Exclusion Criteria:

1. Impossible to walk (wheel chair or bedridden)
2. Diabetic foot
3. Unhealed and/or painful foot injury
4. Acquired deformity of a foot (osteophytosis, parrot beak on metatarso-phalangeal joint of the first ray, a bunion or hallux valgus, or hallux rigidus or stiffness of the big toe)
5. Intercurrent disease that may interfere with the evaluation of the primary outcome (Parkinson's disease, peripheral neuropathy, Little's disease, significant hip or knee injury)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Difference in timed walking performance for 30 steps on the pathological side between D0 and D30. | Day 30